CLINICAL TRIAL: NCT07112469
Title: Physical Activity and Sleep Time Per Day of Junior High School Students in Ho Chi Minh City and the Effectiveness of Interventions to Increase Physical Activity and Sleep Time
Brief Title: The Effectiveness of Intervention to Increase Physical Activity and Sleep Time of Junior High School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pham Ngoc Thach University of Medicine (Other)
Responsible Party: Principal Investigator, Hong Tang, Vice Dean of the Faculty of Public Health, Pham Ngoc Thach University of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4682/QĐ-ĐHYD
Record Dates: First submitted 2025-07-16; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Moderate Physical Activity (MPA); Vigorous Physical Activity (VPA); Moderate to Vigorous Physical Activity (MVPA); Total of Sleep Time (TST)
Keywords: physical activity; sleep time; junior school students; Ho Chi Minh city; intervention
MeSH Terms: conditions — Motor Activity | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: Cross-sectional survey study among 948 students in grades 6 to 9, from 12 secondary schools in Ho Chi Minh City to describe personal characteristics and family factors of students; exercise and sleep environment, identify factors related to MVPA time and TST. In the intervention phase, the investigators selected 8 schools from 12 schools, including 4 schools as the intervention group and 4 schools as the control group. Then, the investigators evaluated the effectiveness of the intervention by increasing MVPA time and TST after 1 month and 6 months between the two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental): The intervention group students were selected as follows: from the 12 participating schools in Phase 1, 8 clusters (where each cluster was a school) were randomly selected. From these 8 schools, 4 were randomly assigned to the intervention group and 4 to the control group. The students selected for intervention were those who had participated in the Phase 1 survey.
  Interventions: Behavioral: Health promotion communication; Behavioral: Guidance and practice in developing physical activity plans
- No intervention group (No Intervention): After randomly selecting a similar cluster of schools as described in the intervention group, students who had participated in the Phase 1 survey were re-surveyed one and six months after the completion of the intervention activities in the intervention group.

INTERVENTIONS:
Behavioral: Health promotion communication — 1. Students (Research subjects):
     * All students: Students perform plays during flag-raising ceremonies for all grades. These plays emphasize the importance of increasing physical activity for better health.
     * Selected students from Phase 1: Students selected in Phase 1 are guided to play games that help them identify healthy behaviors. They also receive flyers with messages about the benefits of physical activity.
  2. Parents:
     Parents receive flyers with messages about the benefits of physical activity.
  3. Schools:
  Research team advises school principals and discusses ways to adjust factors that affect students' physical activity time. These factors are assessed based on cross-sectional study results, literature reviews, and the evaluation of the current situation at each school.
  Arms: Intervention group
Behavioral: Guidance and practice in developing physical activity plans — The intervention is exclusively implemented for students who participated in the Phase 1 survey. These students are being guided to create weekly physical activity plans by keeping a journal. They are also encouraged to self-monitor their progress. A Facebook page has been created to launch the "Active Moments with Family" challenge and provide regular health-related updates. Teachers are sharing this page with parents to promote participation in the challenge and enhance their health knowledge.
  Arms: Intervention group

SUMMARY:
The study comprises 2 phases. Phase 1: Cross-sectional study investigated the duration of moderate to vigorous physical activity (MVPA) time and the total of sleep time (TST), describing and identifying factors related to duration of MVPA time and TST. Phase 2: Conduct an intervention to evaluate the effectiveness and factors related to physical activity and sleep time average day of secondary school students in Ho Chi Minh City.

DETAILED DESCRIPTION:
Detailed of 2 phases in this study below:

Phase 1: Cross - sectional study

A cross-sectional study was conducted in 12 schools, with 2 classes selected from each school (one from grades 6-7 and one from grades 8-9). The study included a total of 948 participants with complete data for analysis (achieving the minimum sample size of 942 students). At this phase, objectives were: 1) To determine the average daily duration of MVPA and TST. 2) To investigate the association between MVPA and TST and various factors (student, family, and environmental). The sequence of activities was as follows:

1. Research team contacted the school administration to send research questionnaires and informed consent forms to students and parents of the selected classes.
2. On the survey day, researchers collected consent forms and instructed students to complete a self-management questionnaire about personal characteristics, family background, physical activity environment, and sleep habits. Afterwards, researchers guided consenting students in wearing Actigraph GT9X accelerometers, providing them with log sheets to record daily wear times.
3. After 7 consecutive days of accelerometer wear, the research team returns to the schools to collect the devices from the school health offices. Data from the accelerometers were included in the analysis only if students have worn the device for at least four days, including at least one weekend day.
4. Student physical activity and sleep data extracted using ActiLife software. The extracted parameters included: time spent in moderate-intensity physical activity (MPA), vigorous-intensity physical activity (VPA), moderate-to-vigorous physical activity (MVPA), total sleep time (TST), sleep efficiency (SE), wake after sleep onset (WASO), time in bed (TIB), and number of days with accelerometer wear.
5. Following data extraction and accelerometer recalibration, the research team continues to conduct surveys at the remaining schools as planned until the target sample size is reached.
6. Upon completion of data collection, data from all 12 schools is consolidated into a unified dataset. Response rates are calculated, and data cleaning is conducted. Subsequently, data analysis is performed to meet the objectives of Phase 1.

Phase 2: Interventional study

Students from classes of 8 schools in all 12 participating schools were selected from Phase 1. They were divided into intervention and control groups, each comprising 4 schools. The research team implemented intervention activities in the intervention group and evaluated the intervention's effectiveness after 1 and 6 months in both groups to compare changes. The objectives of Phase 2 included: 1) To compare changes in MVPA duration between the intervention and control groups before and after the intervention; 2) To compare changes in sleep quality between the intervention and control groups before and after the intervention. For the intervention group activities, the research team focused on counseling, health education, and guidance on developing plans to improve physical activity in students. The investigators implemented interventions in the following groups:

1. Students: all students from the 4 schools and students who participated in Phase 1
2. Parents
3. School administrators Besides that, 4 remaining schools in the control group continued their regular academic activities without any additional interventions related to physical activity or sleep.

The researcher assessed the changes in MVPA and sleep quality between the intervention and control groups after 1 and 6 month Actigraph using.

ELIGIBILITY:
Inclusion criteria:

1. For school: All public secondary schools located in the district of Ho Chi Minh city.
2. For student: Students (aged 10 - 16) attending grades 6, 7, 8, and 9 in public secondary schools located in the districts of Ho Chi Minh City.

Exclusion criteria:

1. For school: All public secondary schools located in the district of Ho Chi Minh city. do not cooperate in the research.
2. For student: Students or parents of students do not agreement to participate in the study.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 948 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Average Daily MVPA and TST | From enrollment to the end of intervention at 6 months
  Student MVPA calculations:
  * Accelerometer data was collected to measure students's physical activity. This data was processed using ActiLife software to classify different intensity levels of activity. Subsequently, the time spent in MVPA was analysised. Variables extracted alongside included MPA, VPA.
  * Average daily MVPA was calculated by average of weekdays (5 days) and weekend days (2 days). Unit of MVPA was minutes per day per student. The calculated results were analyzed using cluster analysis, considering the weight of each student in different clusters.
  Student TST calculations:
  Just as MVPA was calculated, sleep data was obtained from accelerometer readings and processed using ActiLife. TST was calculated and adjusted to reflect the full week distribution. Other variables such as TIB, WASO, and SE were also extracted from the dataset. TST is measured in hours per day per student. The calculated results are analyzed using cluster analysis, taking into account the weight.
Changes in MVPA and TST at 1 month and 6 months follow-ups between intervention and control groups | From enrollment to the end of intervention at 6 months
  * After 1 month and 6 month of intervention, the study reassessed students' MVPA and TST using accelerometers and extracted similar information as described in Outcome 1. Paired t-tests were used to compare the intervention and cross-sectional phases to examine the pre-post intervention differences in the intervention group (similarly for the control group).
  * The differences in MVPA and TST between the two groups were compared at 1-month and 6-month follow-ups. It was hypothesized that after 1 month, the intervention group would show an increase in MVPA and TST compared to the cross-sectional phase, while the control group would show no change compared to the baseline. After 6 months of intervention, the intervention group would still show an increase in MVPA and TST compared to the cross-sectional phase, but the increase would be less significant than the 1-month assessment, while the control group would show no change compared to the baseline.

SECONDARY OUTCOMES:
Associations of MVPA and TST with factor groups derived from questionnaire responses | From enrollment to the end of intervention at 6 months
  The variables investigated in Phase 1 through a questionnaire included:
  1. Individual factors: age, gender, grade level, body mass index (BMI), and self-reported physical activity participation.
  2. Family factors: parental occupation, parental physical activity, parental bedtime, family reminder for children's bedtime, and family encouragement for physical activity.
  3. Environmental factors: availability of physical activity facilities in the neighborhood and school environment, and sleep environment characteristics.
  Frequency and proportion for categorical variables: school, class, subgroup, BMI subgroup, qualitative characteristics of family, qualitative characteristics of physical and sleep environments. Mean and standard deviation for normally distributed quantitative variables, and median and interquartile range for non-normally distributed quantitative variables: age, BMI, parental bedtime. Linear regression analysis within cluster analysis will be used to assess the relationshi

CONTACTS AND LOCATIONS:
Locations (1):
- Junior high school, Ho Chi Minh City, Vietnam